CLINICAL TRIAL: NCT07019948
Title: The Correlation Between Sleep Quality and Sleep Aid Use and Dietary Patterns of Medical Staff in Emergency and Critical Care Departments
Brief Title: The Correlation Between Sleep Quality and Sleep Aid Use and Dietary Patterns
Status: Not yet recruiting | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Association Profession, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: K-2024-127-01
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-07

CONDITIONS: Sleep Disorder (Disorder)
Keywords: sleep quality; Sleep disorders; Sedative-hypnotic drugs; Dietary pattern; Clinical medical staff
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Medical staff in emergency and critical department: Medical staff in emergency and critical departments of some tertiary hospitals in Guangzhou. Medical staff who have obtained the qualification certificate of doctors and nurses through practice registration.； Working in the emergency and critical care departments for more than 1 year ； No serious physical disease and psychiatric history； being able to communicate in Chinese.

SUMMARY:
In this study, medical staff in emergency and critical care departments were investigated. It was assumed that the use of sleep aids and dietary patterns affected their sleep quality. The structural equation model was used to analyze the status of sleep quality of medical staff in emergency and critical care departments, and to explore the effects of sleep aids and dietary patterns on sleep quality and its mechanism.

( 1 ) Is the overall sleep quality of medical staff in emergency and critical departments poor ( 2 ) Do medical staff with poor sleep quality in acute and critical departments use sleep aids more frequently ( 3 ) Is there a correlation between sleep quality and certain dietary patterns among medical staff in emergency and critical care departments ( 4 ) Are there significant differences in dietary choices among medical staff in emergency and critical departments using sleep aids

ELIGIBILITY:
Inclusion Criteria:

* Medical staff who have obtained the qualification certificate of doctors and nurses through practice registration
* Working in the emergency and critical care departments for more than 1 year
* No serious physical disease and psychiatric history
* be able to communicate in Chinese

Exclusion Criteria:

* Interns, students or trainees
* The last six consecutive months of sick leave, maternity leave, out of the learner
* Non-night shift workers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical staff in emergency and critical care departments of tertiary hospitals in Guangzhou City
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
sleep quality | baseline
  The Pittsburgh Sleep Quality Index scale is used to measure participants' sleep quality. The total score ranges from 0 to 21. Higher scores indicate lower quality of sleep.
Sedative-hypnotic drugs | baseline
  The questionnaire on the use of sleep medications included whether or not sleep medications were used, the time of the first use of sleep medications, the types of sleep medications used, the frequency of use, the reasons for use, the average amount of each use, the source of sleep medications, the effect of sleep medications, whether the doctor was consulted, whether it was considered that the use of sleep medications would lead to drug dependence, the side effects of the use of sleep medications, the impact of sleep medications on work and life, etc. The purpose is to gain an in-depth understanding of the characteristics of the use of sleep medications in the study subjects.
Food intake | baseline
  In this study, the simplified Chinese food frequency questionnaire was used to divide the food into 19 food groups according to the food category of the ' Chinese food composition table ' : including cereals, grains, potatoes, beans and their products, livestock meat, poultry meat, fish, shrimp, crab, shellfish, fresh eggs, milk and its products, vegetables, fungi and algae, fruits, pickles, fast food, snacks, beverages, tea, wine, coffee. According to whether the intake, the frequency of intake ( times / day, times / week, times / month, times / year ) and the average intake ( g / ml ), the food intake in the last month was asked and converted into daily food intake.

SECONDARY OUTCOMES:
Depression-anxiety-stress situation | baseline
  The Chinese version of the Depression-Anxiety-Stress Scale was used. The three subscales of depression, anxiety and stress each contain 7 items, all of which use a 4-level score from ' 0 ' ( inconsistent ) to ' 3 ' ( always consistent ). The scores of each subscale are multiplied by 2, which is the score of the subscale. The higher the score, the more this emotion is.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia PHD, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No